CLINICAL TRIAL: NCT04961970
Title: Hepatic Arterial Infusion Chemotherapy of Oxaliplatin, 5-Fluorouracil and Leucovorin Versus Systemic Chemotherapy of Gemcitabine and Cisplatin for Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: HAIC With FOLFOX Versus Systemic Chemotherapy With GP for Unresectable ICC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Ming (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S035B
Record Dates: First submitted 2021-07-07; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; systemic chemotherapy; hepatic artery infusion chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatic artery infusion chemotherapy (Experimental): Participants received hepatic artery infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin
  Interventions: Drug: oxaliplatin , fluorouracil, and leucovorin
- Systemic chemotherapy (Active Comparator): Participants received systemic chemotherapy of gemcitabine and cisplatin
  Interventions: Drug: gemcitabine and cisplatin

INTERVENTIONS:
Drug: oxaliplatin , fluorouracil, and leucovorin — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Arms: Hepatic artery infusion chemotherapy
Drug: gemcitabine and cisplatin — administration of gemcitabine and cisplatin via vein
  Arms: Systemic chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin compared systemic chemotherapy of gemcitabine and cisplatin in patients with unresectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ICC
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* Without distant metastasis, but intrahepatic lymph node metastasis is allowed
* The following laboratory parameters:

Platelet count ≥ 50,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/ L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-07-09 (Estimated); Primary Completion 2025-07-09 (Estimated); Study Completion 2025-07-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression free survival | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Time to progression | 12 months
  TTP was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST).
Number of adverse events. | 30 days
  Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China